CLINICAL TRIAL: NCT05917990
Title: Text-Messaging Communication Micro-Intervention for Couples Coping With Advanced GI Cancer
Brief Title: Dyadic Text-Messaging Micro-Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI accepted a faculty position at a different institution, and the postdoctoral grant was terminated
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113252; 1F32CA278417-01 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2023-06-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer; Gastrointestinal Cancer
Keywords: Cancer; Couples
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic Text-Messaging Micro-Intervention (Experimental): The proposed micro-intervention will consist of 4 modules: welcome and overview module, sharing thoughts and feelings module, problem-solving skills module, and meaningful experiences and resources module. Each of the modules contain information and skills relevant to improving dyadic communication and relationship functioning in couples coping with advanced cancer.
  Interventions: Behavioral: Dyadic Text-Messaging Micro-Intervention
- Waitlist Control (No Intervention): Couples in the waitlist control group will not initially receive any intervention materials; after completing post-assessment, couples in this arm will be offered the dyadic micro-intervention.

INTERVENTIONS:
Behavioral: Dyadic Text-Messaging Micro-Intervention — Participants receive text-messages consisting of information and skills relevant to improving couples' communication and relationship functioning.
  Arms: Dyadic Text-Messaging Micro-Intervention

SUMMARY:
The purpose of this study is to develop, refine, and pilot test a text-messaging micro-intervention focused on improving communication skills for couples in which one partner has gastrointestinal cancer.

For the pilot testing portion of the study, couples will be randomized (1:1) to receive the text-messaging communication micro-intervention or to a waitlist control group. All couples will be asked to complete questionnaires before randomization and 30 days post-randomization. Couples in the waitlist control group will be offered the text-messaging micro-intervention after completing the second set of surveys (30-days post-randomization).

DETAILED DESCRIPTION:
A cancer diagnosis requires patients and their intimate partners to communicate effectively to navigate illness-related challenges. Research indicates that couples who use effective communication strategies have better individual psychological adjustment and higher relationship satisfaction. However, many couples have difficulty communicating about cancer-related issues which can lead to poorer individual, relationship, and patient health outcomes.

While dyadic interventions to improve couple communication have proven efficacious, they are often time intensive and have limited reach. The challenges of recruiting couples into dyadic interventions are well-documented, with low recruitment rates especially among underserved couples.

Micro-interventions, which consist of brief educational materials and short activities delivered via text message or a mobile application, have significant potential to increase reach and participation in diverse groups of couples by increasing flexibility and reducing barriers to access. Previous studies have found micro-interventions to be effective in promoting health behavior change in a wide range of individuals and in enhancing dyadic functioning in community couples.

The proposed project aims to develop, test, and examine the feasibility, acceptability, and efficacy of a text-messaging communication micro-intervention for couples coping with advanced GI cancer.

ELIGIBILITY:
Inclusion Criteria:

1. In a committed relationship
2. Both members of the couple must read and speak fluent English
3. One partner must be diagnosed with advanced (Stage III or IV) gastrointestinal cancer and undergoing systemic therapy (e.g., chemotherapy)
4. One or both partners must score ≥1.0 on the holding back screen

Exclusion Criteria:

1. Patient or partner who is unable to provide informed consent as assessed by the oncologist or research staff
2. Patient or partner is physically impaired in such a way that precludes the use of a mobile device
3. Patient or partner who do not have a mobile device
4. Patient or partner who is too sick to participate, as judged by the oncologist or research staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of acceptability of micro-Intervention | Post-Intervention (30 days post randomization)
  Acceptability of treatment will be measured using the Client Satisfaction Questionnaire (CSQ-8); higher scores indicate higher satisfaction
Changes in relationship satisfaction | Baseline (after informed consent, prior to randomization), Post-Intervention (30 days post randomization)
  Changes in relationship satisfaction measured by the Couples Satisfaction Index (CSI-4); higher scores indicate higher relationship satisfaction
Changes in constructive communication | Baseline (after informed consent, prior to randomization), Post-Intervention (30 days post randomization)
  Changes in constructive communication measured by the Communication Patterns Questionnaire (CPQ-Short Form)

CONTACTS AND LOCATIONS:
Overall Officials: Karena Leo, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No